CLINICAL TRIAL: NCT02484001
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) as Monotherapy for Patients With Newly Diagnosed Partial-onset Seizures: a Double-blind, Randomized, Active-controlled, Parallel-group, Multicenter Clinical Study - Open-label ESL Extension
Brief Title: Eslicarbazepine Acetate (BIA 2-093) as Monotherapy in Patients With Newly Diagnosed Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-311/EXT
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Epilepsy
Keywords: Eslicarbazepine acetate; BIA 2-093; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ESL 800 mg (Experimental): ESL will be administered orally once daily (QD)
  Interventions: Drug: ESL 800 mg
- ESL 1200 mg (Experimental): ESL will be administered orally once daily (QD)
  Interventions: Drug: ESL 1200 mg
- ESL 1600 mg (Experimental): ESL will be administered orally once daily (QD)
  Interventions: Drug: ESL 1600 mg
- ESL 400 mg (Experimental): ESL will be administered orally once daily (QD)
  Interventions: Drug: ESL 400 mg

INTERVENTIONS:
Drug: ESL 800 mg — one (1) tablet of 800 mg (QD).
  Other Names: BIA 2-093
  Arms: ESL 800 mg
Drug: ESL 1200 mg — one (1) and a half tablets of 800 mg (QD). ESL tablets are scored and can be divided in two equal halves (each one containing 400 mg ESL)
  Other Names: BIA 2-093
  Arms: ESL 1200 mg
Drug: ESL 1600 mg — two (2) tablets of 800 mg (QD).
  Other Names: BIA 2-093
  Arms: ESL 1600 mg
Drug: ESL 400 mg — half tablet of 800 mg (QD). ESL tablets are scored and can be divided in two equal halves (each one containing 400 mg ESL)
  Other Names: BIA 2-093
  Arms: ESL 400 mg

SUMMARY:
This is a Phase III, multinational, open-label, non-controlled study with subjects under treatment in the double-blind BIA-2093-311 study (NCT01162460).

Subjects will enter the open-label extension study after the preceding double-blind study was unblinded and they are attending their last Extension Phase Visit (EPV) of the double-blind study.

For all subjects, the day of the last EPV of the double-blind study will also be the day of Visit 1 for the open-label extension study. All subjects will receive Eslicarbazepine acetate (ESL) under open-label conditions at Visit 1.

The complete study duration including treatment with ESL under open-label conditions and follow-up is expected to last approximately 2 years (105 weeks).

In case ESL as monotherapy will achieve MA prior to the end of 2017, the study may be discontinued prematurely within 42 days after achievement of MA.

DETAILED DESCRIPTION:
For all subjects participating in this open-label extension study, the last Extension Phase Visit (EPV) of the double-blind study will also be the day of Visit 1 for this study. At this visit, the subjects will be asked if they are willing to continue in an open-label extension and to receive treatment with Eslicarbazepine acetate (ESL) for up to additional 2 years. In case marketing authorization (MA) of ESL as monotherapy will be achieved prior to the end of 2017, the study may be discontinued prematurely within 42 days after achievement of MA.

For subjects not willing to enter the extension study, IMP from the double-blind study (CBZ-CR or ESL) is to be discontinued according to the down-titration scheme in the clinical study protocol and commercially available antiepileptic drug (AED) is to be introduced according to investigator's discretion.

In case the subject is willing to enter the extension study, subjects already treated with ESL will continue with their last evaluated dose (ESL 800 mg, 1200 mg or 1600 mg QD).

Subjects previously treated with CBZ-CR will start with ESL 400 mg QD for one week followed by up-titration to the ESL target dose which is equivalent to the last evaluated CBZ-CR dose level (i.e. CBZ-CR 200 mg BID -> ESL 800 mg QD; CBZ-CR 400 mg BID -> ESL 1200 mg QD; CBZ-CR 600 mg BID -> ESL 1600 mg QD) in steps of 400 mg dose increase per week.

All subjects previously treated with CBZ-CR, regardless of their last evaluated dose level, will start CBZ-CR down-titration two weeks after first receipt of ESL treatment as part of the double-blind study and as outlined in the BIA-2093-311 study protocol.

In case of new seizures, the ESL dose can be increased to a maximum dose of ESL 1600 mg QD [dose level C], depending on the investigator's decision. Any up-titration should be performed in weekly steps of 400 mg.

If according to the investigator's opinion the subject may benefit from a combination treatment, an additional commercially available AED as add-on can be introduced at the investigator's discretion.

If deemed necessary by the investigator, e.g. due to occurrence of adverse events, the dose of ESL can be reduced according to investigator's discretion, as long as the dose remains in the range of 800 mg QD to 1600mg QD.

In case the subject started with the extension study but is not willing to continue at any time, the subject has to be switched to commercially available AEDs to receive the best standard of care according to the investigator's discretion. Down-titration of ESL as required should be performed in steps of 400 mg decrease per week

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the extension study, subjects must fulfill all of the following at Visit 1 (Day 1, start of the open-label extension study):

1. Participated in the preceding double-blind study and were still ongoing at the time of unblinding.
2. Have signed informed consent before undergoing any activities related to the open-label extension study.
3. Demonstrated cooperation and willingness to complete all aspects of the study.
4. Female subjects without childbearing potential (2 years postmenopausal, bilateral oophorectomy or tubal ligation, or complete hysterectomy) are eligible. Female subjects with childbearing potential must not be pregnant as confirmed by a negative serum ß-human chorionic gonadotropin (hCG) test and sexually active females must be using a medically acceptable effective non-hormonal method of contraception for the duration of the study and until the Post-study Visit (PSV).

Exclusion Criteria:

Subjects having any of the following at Visit 1 are to be excluded from the study:

1. Excluded from the double-blind study due to seizure in the Maintenance or Extension Phase, or at dose level C (either CBZ-CR or ESL), or discontinued prematurely due to any other reason in the double-blind study.
2. Presence of any major protocol violation during the double-blind study which may have an impact on the compliance during this extension study.
3. Judged clinically to have a suicidal risk in the opinion of the investigator based upon a clinical interview and the Columbia Suicide-Severity Rating Scale (C-SSRS).
4. Occurrence of an adverse event (AE) indicating a suspected presence of atrioventricular block (2nd degree and above) or of any other AEs during the double-blind study which are judged by the investigator as contraindicative to further participation in the open-label extension study.
5. Events of alcohol, drug, or medication abuse during the preceding double-blind study.
6. Relevant clinical laboratory abnormalities (e.g. sodium <125 mmol/L, alanine or aspartate transaminases >2 x the upper limit of normal, white blood cell count <3000 cells/mm3) (as reported at Visit 1).
7. Pregnancy or lactating.
8. Any other condition or circumstance that, in the opinion of the investigator, could compromise the subject's ability to comply with the extension-study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | up to 2 years
  Time to treatment failure, defined as time from start of open-label ESL treatment at Visit 1 until withdrawal due to AE or due to lack of efficacy (i.e. inadequate seizure control), is the primary endpoint of this study. Open-label ESL treatment will be provided for approximately 2 years. Regular Treatment Visits (TVs) will be performed every 3 months after start of treatment.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) reported by patient | participants will be followed for the duration of the clinical trial, an expected average of 2 years
  The investigator will monitor AEs at each visit, from signing of informed consent throughout the study, including at Early Discontinuation Visit (EDV), End-of-study (EOS) Visit, and Post-study Visit (PSV), using an unstructured interview and by review of the subject diaries. The investigator will inquire generally about the subject's well-being since the last visit. Details of any reported AEs will be recorded at all scheduled and unscheduled visits as well as those reported during any telephone contact. In addition, comments in the subject diaries will be reviewed by the investigator and any events considered by the investigator to be an AE will be recorded as such.

REFERENCES:
- [Derived] Trinka E, Rocamora R, Chaves J, Koepp MJ, Ruegg S, Holtkamp M, Moreira J, Fonseca MM, Castilla-Fernandez G, Ikedo F. Lipid profile with eslicarbazepine acetate and carbamazepine monotherapy in adult patients with newly diagnosed focal seizures: post hoc analysis of a phase III trial and open-label extension study. Ther Adv Neurol Disord. 2023 Sep 4;16:17562864231193530. doi: 10.1177/17562864231193530. eCollection 2023. PMID 37675038